CLINICAL TRIAL: NCT03577964
Title: Development of Pneumonia Due to Alveolar Glucose Levels in Systemic Hyperglycemia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Robert Kraft MD, MMS, Pricipal Investigator of Clinical Research, Dept of Cardiac, Thoracic and Vascular Surgery, University of Ulm
Other Study IDs: 267/17
Record Dates: First submitted 2018-06-07; First posted 2018-07-05 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Glucose Metabolism Disorders; Pneumonia, Bacterial
Keywords: Pneumonia; Glucose; Infections; Respiratory Tract Infection; Hyperglycemia; Critical Care
MeSH Terms: conditions — Glucose Metabolism Disorders; Pneumonia, Bacterial; Pneumonia; Infections; Respiratory Tract Infections; Hyperglycemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Glucose Measurements, — Measurement of glucose Levels in bronchio alveolar secretions

SUMMARY:
Incidence of Pneumonia in Patients with high systemic glucose levels.

DETAILED DESCRIPTION:
Clinical and mechanistic studies have shown that a hyperglycaemic metabolic condition is associated with a higher incidence of infection and consecutive increased morbidity and mortality. The underlying mechanisms in detail are not completely understood. So far it is not clear whether systemic increased glucose levels are caused by a stress reaction of the body through a catabolic metabolism situation as well as a "stress-induced insulin resistance", or infections are promoted by hyperglycemia. From in vivo and in vitro studies, a glucose threshold for the lung is known (147 mg / dL), similar to that in the kidney. It can be hypothesized, that an intra-alveolar glucose in turn promotes bacterial growth as a nutrient substrate. The aim of the study is to determine the concentration of glucose in the alveolar space in connection with hyperglycemic conditions, and to demonstrate a higher incidence of pneumonia in this patient group. The study will enroll cardiac surgery patients receiving surgical treatment and expected postoperative ventilation. Systemic blood glucose monitoring is recorded throughout hospitalization, as well as the removal of bronchial aspirates intraoperatively and during ventilation to measure glucose levels and bacterial levels. The incidence of pneumonia is recorded during the postoperative period by means of radiological examinations and / or microbiological examinations.

ELIGIBILITY:
Inclusion Criteria:

* women and men over the age of 18 years
* voluntary consent to study participation of the patient
* Planned cardiac surgery with expected endotracheal ventilation of ≥ 1 day postoperatively

Exclusion Criteria:

* age <18 years
* pregnancy
* Non-able-bodied patients (disempowerment / loss of consciousness, limitation of the ability to express one's own will, for example through disability)
* subsequently withdrawn consent
* accommodation in an institution on the basis of official or court orders
* lack of or insufficient knowledge of German language, whereby the understanding of the written patient education is not guaranteed.
* Immunosuppressed patients
* Patients with a malignant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving an planned cardiac surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2020-04-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of pneumonia or lower respiratory tract infection | 20 days post surgery
  The incidence of pneumonia or lower respiratory tract infection will be determined by chest x-ray, CT-Scan and/or sampling of specimens of the lower tract of the airways.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kraft, MD, MMS, Principal Investigator — University of Ulm Dept. of Cardiothoracic and Vascular Surgery
Locations (1):
- University of Ulm Dept. of Surgery, Ulm, Baden Wüttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kraft R, Herndon DN, Mlcak RP, Finnerty CC, Cox RA, Williams FN, Jeschke MG. Bacterial respiratory tract infections are promoted by systemic hyperglycemia after severe burn injury in pediatric patients. Burns. 2014 May;40(3):428-35. doi: 10.1016/j.burns.2013.07.007. Epub 2013 Sep 25. PMID 24074819
- [Background] Wood DM, Brennan AL, Philips BJ, Baker EH. Effect of hyperglycaemia on glucose concentration of human nasal secretions. Clin Sci (Lond). 2004 May;106(5):527-33. doi: 10.1042/CS20030333. PMID 14678009
- [Background] Kalsi KK, Baker EH, Fraser O, Chung YL, Mace OJ, Tarelli E, Philips BJ, Baines DL. Glucose homeostasis across human airway epithelial cell monolayers: role of diffusion, transport and metabolism. Pflugers Arch. 2009 Mar;457(5):1061-70. doi: 10.1007/s00424-008-0576-4. Epub 2008 Sep 10. PMID 18781323
- [Background] Philips BJ, Redman J, Brennan A, Wood D, Holliman R, Baines D, Baker EH. Glucose in bronchial aspirates increases the risk of respiratory MRSA in intubated patients. Thorax. 2005 Sep;60(9):761-4. doi: 10.1136/thx.2004.035766. PMID 16135681

DOCUMENTS (2):
  • Study Protocol (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT03577964/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT03577964/SAP_001.pdf